CLINICAL TRIAL: NCT02235961
Title: A First Human Dose Trial Investigating Safety, Tolerability and Pharmacokinetics for Single Doses of NNC9204-0530 Alone and in Combination With Liraglutide in Overweight to Obese But Otherwise Healthy Male Subjects.
Brief Title: Investigate Safety, Tolerability and Pharmacokinetics for Single Doses of NNC9204-0530 Alone and in Combination With Liraglutide in Overweight to Obese But Otherwise Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9030-4111; U1111-1151-0761 (Registry Identifier: WHO)
Record Dates: First submitted 2014-09-02; First posted 2014-09-10 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Experimental)
  Interventions: Drug: NNC9204-0530; Drug: placebo
- Part 2 (Experimental)
  Interventions: Drug: NNC9204-0530; Drug: liraglutide; Drug: placebo

INTERVENTIONS:
Drug: NNC9204-0530 — Administered as single subcutaneous (s.c., under the skin) injections.
Drug: liraglutide — Administered as subcutaneous (s.c., under the skin) injections of 1.8 or 3.0 mg.
  Arms: Part 2
Drug: placebo — Administered as single subcutaneous (s.c., under the skin) injections.

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of the trial is to investigate safety, tolerability and pharmacokinetics (the exposure of the trial drug in the body) for single doses of NNC9204-0530 alone and in combination with liraglutide in overweight to obese but otherwise healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male, age between (both inclusive) 18 and 55 years at the time of signing inform consent
* Overweight or obese but otherwise healthy male subjects; BMI of between or equal to 27.0 and 35.0 kg/m^2

Exclusion Criteria:

* Thyroid stimulating hormone values outside 0.4-6.0 mIU/l
* HbA1c (glycated hemoglobin) above or equal to 6.5%
* Any clinically relevant ECG (electrocardiogram) findings (e.g. 2nd or 3rd degree AV-block), in particular subjects with repeated demonstration of a QTcF (QT interval corrected by Fridericia formula) interval above 430 ms
* A history of additional risk factors for Torsades de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* The use of concomitant medications that prolong the QT/QTc interval
* Obesity caused by endocrinology disorders (e.g. Cushing's Syndrome)
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2
* Calcitonin above 50 ng/L
* History of pancreatitis (acute or chronic)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 2014-09-04 (Actual); Primary Completion 2016-07-06 (Actual); Study Completion 2016-07-06 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events recorded | From time of dosing of NNC9204-0530 (Day 1) until completion of the follow-up visit (Day 21-27)

SECONDARY OUTCOMES:
Area under the NNC9204-0530 serum concentration-time curve | From dosing visit to infinity calculated on 0-24 days NNC9204-0530 serum concentration-curve based on 21 sampling points
Maximum concentration of NNC9204-0530 in serum | From dosing visit to infinity calculated on 0-24 days NNC9204-0530 serum concentration-curve based on 21 sampling points
The time to maximum concentration of NNC9204-0530 in serum | From dosing visit to infinity calculated on 0-24 days NNC9204-0530 serum concentration-curve based on 21 sampling points
The terminal half-life of NNC9204-0530 | From dosing visit to infinity calculated on 0-24 days NNC9204-0530 serum concentration-curve based on 21 sampling points

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com